CLINICAL TRIAL: NCT05708924
Title: MT2021-27 Intraperitoneal FT538 With Intravenous Enoblituzumab in Recurrent Ovarian, Fallopian Tube, and Primary Peritoneal Cancer
Brief Title: MT2021-27 FT538 Recurrent Ovarian, Fallopian Tube, and Primary Peritoneal Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Product withdrawn from clinical development
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2021LS103; P01CA111412 (NIH)
Record Dates: First submitted 2022-12-14; First posted 2023-02-01 (Actual); Results first posted 2025-08-14 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-07

CONDITIONS: Cancer; Solid Tumor; Ovarian Cancer; Peritoneal Cancer; Fallopian Tube Cancer
MeSH Terms: conditions — Neoplasms; Ovarian Neoplasms; Fallopian Tube Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- IP FT538 monotherapy (Experimental): Level -1: IP FT538 monotherapy 5 x 10^7 cells/dose Level 1: IP FT538 monotherapy 1 x 10^8 cells/dose Level 2: IP FT538 monotherapy 3 x 10^8 cells/dose Level 3: IP FT538 monotherapy 1 x 10^9 cells/dose Level 4: IP FT538 monotherapy 1.5 x 10^9 cells/dose
  Interventions: Drug: FT538
- IP FT538 + Enoblituzumab (Experimental): Level 5: IP FT538 at the safe dose (MTD-1) + Enoblituzumab Level 6: IP FT538 at the highest dose (MTD) + Enoblituzumab
  Interventions: Drug: FT538; Biological: Enoblituzumab

INTERVENTIONS:
Drug: FT538 — FT538 IP at assigned dose level on Day 1, Day 8, and Day 15.
Biological: Enoblituzumab — Enoblituzumab 15 mg/kg IV begin on Day -6 and continuing once every 3 weeks beginning on Day 22 until disease progression or unacceptable toxicity - refer to Section 7.2.1 for timing of the enoblituzumab dose on Day 22 if steroid pre-meds are needed due to an infusion reaction with the 1st enoblituzumab dose as there is a 14 day ban on corticosteroid use after the last dose of FT538
  Other Names: RES242; MGA271
  Arms: IP FT538 + Enoblituzumab

SUMMARY:
To determine the maximum tolerated dose (MTD) of FT538 monotherapy when administered via intraperitoneal (IP) catheter and in combination with intravenous (IV) enoblituzumab in patients with recurrent ovarian, fallopian tube, and primary peritoneal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Recurrent epithelial ovarian cancer, fallopian tube, or primary peritoneal cancer meeting one of the following minimal prior treatment requirements (no limit to the maximum number of prior treatments).
* Platinum Resistant: may receive FT538 as 2nd line (as 1st salvage therapy).
* At least 18 years of age at the time of consent.
* GOG Performance Status 0, 1, or 2 (refer to Appendix I).
* Adequate organ function within 14 days (28 days for pulmonary and cardiac) of study treatment (CY/Flu or enoblituzumab) start
* Pulmonary Function: Oxygen saturation ≥ 90% on room air; PFTs are performed only if known history or as medically indicated - if done, must have pulmonary function >50% corrected DLCO and FEV1.
* Cardiac Function: LVEF ≥ 40% by echocardiography, MUGA, or cardiac MRI; no clinically significant cardiovascular disease including any of the following: stroke or myocardial infarction within 6 months prior to first study treatment; unstable angina or congestive heart failure of New York Heart Association (NYHA) Grade 2 or higher (Appendix I).

Exclusion Criteria:

* Pregnant or breastfeeding or planning on becoming pregnant in the next 6 months.
* Currently receiving or likely to require systemic immunosuppressive therapy
* Active autoimmune disease requiring systemic immunosuppressive therapy.
* History of severe asthma and currently on chronic systemic medications.
* Uncontrolled bacterial, fungal or viral infections with progression of clinical symptoms despite therapy.
* Receipt of any biological therapy, chemotherapy, or radiation therapy (except palliative RT), within 2 weeks prior to the first dose of FT538
* Live vaccine within 6 weeks prior to start of lympho-conditioning.
* Known allergy to the following FT538 components: albumin (human) or dimethyl sulfoxide (DMSO).
* Prior enoblituzumab.
* Non-malignant CNS disease such as stroke, epilepsy, CNS vasculitis, or neurodegenerative disease or receipt of medications for these conditions in the 2-year period leading up to study enrollment. (Refer to Section 5.1.8 regarding history of brain metastases.)
* Known history of HIV positivity or active hepatitis C or B - chronic asymptomatic viral hepatitis is allowed.
* Presence of any medical or social issues that are likely to interfere with study conduct or may cause increased risk to patient.
* Any medical condition or clinical laboratory abnormality that, per investigator judgement, precludes safe participation in and completion of the study or that could affect compliance with protocol conduct or interpretation of results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2023-04-28 (Actual); Primary Completion 2024-08-06 (Actual); Study Completion 2024-08-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Masonic Cancer Center - University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | IP FT538 Monotherapy | IP FT538 + Enoblituzumab
Started | 1 | 0
Completed | 1 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Trial was terminated. Only one participant consented to the study prior to termination.
Groups:
- Total: Total of all reporting groups
Arm/Group | IP FT538 Monotherapy | IP FT538 + Enoblituzumab | Total
Number analyzed (Participants) | 1 | 0 | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 |  | 0
  Between 18 and 65 years | 1 |  | 1
  >=65 years | 0 |  | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 |  | 1
  Male | 0 |  | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 |  | 0
  Not Hispanic or Latino | 1 |  | 1
  Unknown or Not Reported | 0 |  | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  | 0
  Asian | 0 |  | 0
  Native Hawaiian or Other Pacific Islander | 0 |  | 0
  Black or African American | 0 |  | 0
  White | 1 |  | 1
  More than one race | 0 |  | 0
  Unknown or Not Reported | 0 |  | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 |  | 1

OUTCOME MEASURES:

1. Primary Outcome: Determine Maximum Tolerated Dose (MTD) of FT538
Description: The primary objective of the study is to determine the maximum tolerated dose (MTD) of FT538 monotherapy when administered via intraperitoneal (IP) catheter and in combination with intravenous (IV) enoblituzumab in patients with recurrent ovarian, fallopian tube, and primary peritoneal cancer.
  Monitor the patient for signs of acute infusion related reaction during and after IP infusion. For IV infusion signs of a possible reaction are rigors and chills, rash, urticaria, hypotension, dyspnea, and angioedema.
Time Frame: 48 months
Population: Trial was terminated before the outcome measure data were collected.
Arm/Group | IP FT538 Monotherapy | IP FT538 + Enoblituzumab
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Overall Response Rate (ORR)
Description: Overall response rate is defined as number of patients who have a partial or complete response to therapy divided by the total number of patients who received treatment.
Time Frame: 72 months
Population: Trial was terminated before the outcome measure data were collected.
Arm/Group | IP FT538 Monotherapy | IP FT538 + Enoblituzumab
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Determine Progression-free Survival (PFS)
Description: Number of participants experiencing progression free survival at one year follow up
Time Frame: 72 months
Population: Trial was terminated before the outcome measure data were collected.
Arm/Group | IP FT538 Monotherapy | IP FT538 + Enoblituzumab
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Adverse Events
Description: Number of participants experiencing adverse events with the combination of Enoblituzumab and FT538
Time Frame: 72 months
Population: Trial was terminated before the outcome measure data were collected.
Arm/Group | IP FT538 Monotherapy | IP FT538 + Enoblituzumab
Number analyzed (Participants) | 0 | 0

5. Other Pre Specified Outcome: Tumor Biopsies (if Feasible) at the Time of Catheter Placement and Catheter Removal for Study Related Analysis
Description: Tumors will be biopsied to assess tumor microenvironment.
Time Frame: 72 months
Population: Trial was terminated before the outcome measure data were collected.
Arm/Group | IP FT538 Monotherapy | IP FT538 + Enoblituzumab
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 month
Description: No participants enrolled onto IP FT538 + Enoblituzumab arm.
Arm/Group | IP FT538 Monotherapy | IP FT538 + Enoblituzumab
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/0
Other Adverse Events (participants affected / at risk) | 1/1 | 0/0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IP FT538 Monotherapy (N=1) | IP FT538 + Enoblituzumab (N=0)
Anemia (Blood and lymphatic system disorders) | 1 (4) | NA
Lymphocyte count decreased (Investigations) | 1 (5) | NA
Neutrophil count decreased (Investigations) | 1 (3) | NA
White blood cell decreased (Investigations) | 1 (9) | NA
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1) | NA
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | NA
Buttock pain (Musculoskeletal and connective tissue disorders) | 1 (3) | NA
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-09-09): https://cdn.clinicaltrials.gov/large-docs/24/NCT05708924/Prot_SAP_000.pdf
  • Informed Consent Form (2023-10-13): https://cdn.clinicaltrials.gov/large-docs/24/NCT05708924/ICF_001.pdf